CLINICAL TRIAL: NCT06541275
Title: Assessment of the Dynamic Reduction in Volume and Prolonged Shrinkage of Giant and Symptomatic Cerebral Aneurysms Following Combined Endovascular Interventions
Brief Title: Reduction in Volume and Prolonged Shrinkage of Brain Aneurysms After Combined Endovascular Interventions
Status: Enrolling by invitation | Type: Observational
Sponsor: National Centre for Neurosurgery, Republic of Kazakhstan (Other)
Responsible Party: Principal Investigator, Karashash Menlibayeva, Head of the Hospital Management Department, National Centre for Neurosurgery, Republic of Kazakhstan
Other Study IDs: 20240718-03
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Brain Aneurysm
Keywords: brain aneurysm; endovascular flow diverters; neurovascular
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: brain MRI and CT — The diagnostic tests will be conducted at 6, 12, and 24 months of follow-up.

SUMMARY:
The goal of this observational study is to learn about the long-term effects of combined endovascular interventions in participants over the age of 18 who take endovascular interventions employing endoluminal flow diverter stents, with or without coils, and a hybrid approach of combining bypass anastomosis and parent artery occlusion using the endovascular method to treat their giant symptomatic intracranial aneurysms. The main question it aims to answer is:

• How does the methods of endovascular intervention chosen affect the value of the aneurysmal sac shrinkage and volume reduction? Participants underwent endovascular intervention at the hospital will be recruited with further follow-up of 6, 12, and 24 months.

DETAILED DESCRIPTION:
Large (with a diameter of ≥15 mm) and giant (with a diameter of ≥25 mm) intracranial aneurysms represent a distinct subset within the spectrum of cerebral aneurysms, necessitating intricate treatment considerations given their challenging nature and unfavorable natural course. Traditionally characterized by gradual enlargement, these aneurysms frequently progress to rupture, leading to substantial morbidity and higher mortality rates. Additionally, these aneurysms commonly induce peri-aneurysmal edematous changes in the neighboring brain regions. This impact extends to cranial nerves, potentially resulting in functional compromise due to compression of the surrounding brain tissue. The degree of functional impairment is contingent upon the distribution of the cranial nerves within the cerebral circulation.Current treatment options for large and giant cerebral aneurysms involve endovascular interventions employing endoluminal flow diverter stents, with or without coils, and a hybrid approach of combining bypass anastomosis and parent artery occlusion using the endovascular method. These methods have consistently demonstrated high rates of complete aneurysm occlusion and maintain an acceptable safety profile.

2. Previous studies at the National Centre for Neurosurgery. "Management of giant internal carotid aneurysm by extracranial-intracranial bypass and flow diverter stent" and "Early and midterm results of treatment of giant internal carotid artery paraclinoid aneurysms with trapping and flow diverters" has previously been studied and published. The studies included patients who underwent treatment at the Vascular and Functional Neurosurgery Department, National Centre for Neurosurgery, Astana, Kazakhstan.

3. Research Gap and Novelty of a Research Project. Despite the favorable outcomes observed with treatment methods such as endovascular interventions employing endoluminal flow diverter stents, either with or without coils, and a hybrid approach involving bypass anastomosis and parent artery occlusion using the endovascular method, there is a notable lack of comprehensive data on aneurysmal sac shrinkage and complete obliteration rates following these treatments. To address this gap, this study will evaluate the treatment effects specifically on aneurysmal sac shrinkage and volume reduction - crucial factors for a comprehensive assessment of the effectiveness of these interventions.

In parallel, other studies have delved into investigating aneurysm shrinkage following the use of flow diverters with and without coils. Nevertheless, it is crucial to emphasize that these studies failed to take into account the extent of aneurysm closure evaluated using the Raymond Roy scale, as well as data on the deployment of stents assessed using the O'Kelly-Marotta grading system. Additionally, most of the publications are limited to case descriptions only. Notably, these cases did not include an examination of the packing density of the aneurysm. Furthermore, there is a lack of evidence regarding the role of inflammatory factors in the reduction of brain aneurysms following the deployment of flow diverters. In contrast, studies on patients with abdominal aortic aneurysms have explored the influence of preoperative inflammatory markers, such as Neutrophil-to-Lymphocyte (NLR) and Platelet-to-Lymphocyte (PLR) ratios, on post-endovascular aneurysm repair (EVAR) sac shrinkage. These studies have underscored the substantial impact of these inflammatory markers on aneurysm shrinkage following stent placement. Consequently, this prompts consideration for potential research on these variables in cerebral vascular aneurysm model studies.

In summary, while the flow-diverter treatment process typically spans 6 months to a year with the objective of complete aneurysm elimination, there remains a significant lack of data regarding the extended clinical outcomes of flow-diverter therapy, particularly in the context of large-thrombosed aneurysms.

Study Design. Combined Retrospective-Prospective Study.

Primary Objectives. This study will assess the dynamic reduction in volume and prolonged shrinkage of giant and symptomatic cerebral aneurysms following endovascular interventions employing endoluminal flow diverter stents, with or without coils, and a hybrid approach of combining bypass anastomosis and parent artery occlusion using the endovascular methods.

Objectives:

1. Patient Group Formation:

   Retrospective study:

   - analyze the medical records and form a database for further follow-up.

   Prospective study:
   * Form a group of patients who meet the inclusion criteria.
   * Conduct/study MRI/CT, cerebral angiography, and endovascular techniques to confirm the large and giant intracranial aneurysms.
2. Analyze the results:

   * Conduct a detailed analysis and interpretation of the results obtained from selective cerebral angiography and MRA post-surgery.
   * Follow-up every 6 to 12 months.
   * In the endovascular group, categorize aneurysm occlusion using the O'Kelly-Marotta (OKM) grading scale during the procedure.
3. Long-term Outcome Study:

   * Study the long-term results for patients who underwent surgical intervention.
   * Identify factors influencing aneurysmal sac shrinkage and volume reduction.
   * Examine clinical outcomes, considering the type and volume of the surgical intervention.
4. Criteria Development:

   * Develop criteria for selecting the most appropriate type of surgical intervention for patients with large and giant aneurysms.
   * Improve overall treatment efficacy and enhance surgical outcomes based on comprehensive evaluations and long-term observations.

Patietn Safety. The treatment of patients is performed in a hospital accredited by the Joint Commission International by certified neurosurgeons, and using FDA-approved intraoperative devices. The hospital strictly adheres to all national treatment protocols.

Statistical Method. Excel (Microsoft Office) will be used for cleaning and coding the data. Statistical analysis will be performed on Stata statistical software (Stata Corp.). Descriptive data analysis will include reporting of frequencies and/or percentages where applicable. The normal distribution of continuous data will be checked using histograms and scatter plots. Normally distributed continuous variables will be presented as means ± SD, categorical variables will be presented as percentages. Appropriate statistical tests will be used depending on the variables and sample. Outcomes will be tested for association between continuous and categorical variables with Student's t-test, and/or one-way analysis of variance (ANOVA), and/or Wilcoxon signed-rank test, where appropriate. Chi-square test will be used for categorical variables. A p-value of less than 0.05 will be considered statistically significant. Further statistics will be applied where appropriate.

Sample size: The number of patients with a diagnosis of "large and giant intracranial aneurysms" admitted to the Department of Vascular and Functional Neurosurgery at the National Centre for Neurosurgery and underwent endovascular intervention is approximately 15 patients per year. The sample for the retrospective study will be approximately 75 patients. For the prospective study, the sample size calculation with a 95% confidence interval and a power value of 80% resulted in a total of 22 patients. The required sample size will be increased to 27 to account for a potential 20% failure rate in follow-up lost participants. Sample size calculations have been done using OpenEpi.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years and older;
* Participants with large and giant intracranial aneurysms and underwent endovascular interventions within the last 5 years (2019-2023).

Exclusion Criteria:

* Participants under the age of 18;
* Participants with small intracranial aneurysms in the anamnesis and underwent microsurgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population involves participants who were treated at the Vascular and Functional Neurosurgery Department of the National Centre for Neurosurgery in Astana, Kazahstan.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
A value of the aneurysmal sac shrinkage and volume reduction | From enrollment to the further follow-up of 6, 12, and 24 months.
  A detailed analysis and interpretation of the results obtained from selective cerebral angiography and MRA post-surgery at 6, 12, and 24 months will be performed on participants who underwent endovascular interventions for giant symptomatic brain aneurysms. The analysis will assess the dynamic volume reduction and sac shrinkage.

CONTACTS AND LOCATIONS:
Locations (1):
- National Centre for Neurosurgery, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided
The researchers have not yet decided whether all IPD collected throughout the trial or only the IPD used in the results publication will be shared. Additionally, there is no URL available to share the results at this moment.

REFERENCES:
- [Result] Pasqui E, de Donato G, Molino C, Abu Leil M, Anzaldi MG, Galzerano G, Palasciano G. Residual Aneurysmal Sac Shrinkage Post-Endovascular Aneurysm Repair: The Role of Preoperative Inflammatory Markers. Biomedicines. 2023 Jul 6;11(7):1920. doi: 10.3390/biomedicines11071920. PMID 37509562
- [Result] Mitsui T, Nakagawa I, Kotsugi M, Park H, Yokoyama S, Myouchin K, Nakase H. Remarkable shrinkage of a thrombosed giant aneurysm by stent-assisted jam-packed coil embolization. Surg Neurol Int. 2021 Jul 6;12:328. doi: 10.25259/SNI_511_2021. eCollection 2021. PMID 34345469
- [Result] Akiyama R, Ishii A, Kikuchi T, Okawa M, Yamao Y, Abekura Y, Ono I, Sasaki N, Tsuji H, Matsukawa S, Miyamoto S. Predictors of aneurysm shrinkage after flow diversion treatment for internal carotid artery aneurysms: quantitative volume analysis with MRI. Front Neurol. 2023 Dec 21;14:1266460. doi: 10.3389/fneur.2023.1266460. eCollection 2023. PMID 38187156
- [Result] Makhambetov Y, Kaliyev A, Kikuta KI, Smagulov F, Medetov Y, Kulmirzayev M, Kerimbayev T, Kissamedenov N, Tursynkhan A, Doskaliyev A, Akshulakov S. Early and midterm results of treatment of giant internal carotid artery paraclinoid aneurysms with trapping and flow diverters. Acta Neurochir (Wien). 2019 Sep;161(9):1755-1761. doi: 10.1007/s00701-019-04002-3. Epub 2019 Jul 15. PMID 31309305
- [Result] Kaliyev A, Makhambetov Y, Medetov Y, Kulmirzayev M, Dusembayev S, Nurimanov C, Kunakbayev B, Akshulakov S. Management of giant internal carotid aneurysm by extracranial-intracranial bypass and flow diverter stent. Br J Neurosurg. 2023 Dec;37(6):1893-1897. doi: 10.1080/02688697.2021.1947974. Epub 2021 Jul 8. PMID 34236251
- [Result] Dutta G, Singh D, Jagetia A, Srivastava AK, Singh H, Kumar A. Endovascular management of large and giant intracranial aneurysms: Experience from a tertiary care neurosurgery institute in India. J Cerebrovasc Endovasc Neurosurg. 2021 Jun;23(2):99-107. doi: 10.7461/jcen.2021.E2020.08.008. Epub 2021 May 17. PMID 33993689
- [Result] Lawton MT, Spetzler RF. Surgical management of giant intracranial aneurysms: experience with 171 patients. Clin Neurosurg. 1995;42:245-66. PMID 8846596
- [Result] Moon E, Park W, Song Y, Lee DH, Ahn JS, Park JC. Mass Effect After Flow Diversion for Unruptured Large and Giant Cavernous or Paraclinoid Internal Carotid Artery Aneurysm. World Neurosurg. 2023 Dec;180:e108-e116. doi: 10.1016/j.wneu.2023.08.129. Epub 2023 Sep 9. PMID 37690582
- [Result] Lonjon M, Pennes F, Sedat J, Bataille B. Epidemiology, genetic, natural history and clinical presentation of giant cerebral aneurysms. Neurochirurgie. 2015 Dec;61(6):361-5. doi: 10.1016/j.neuchi.2015.08.003. Epub 2015 Dec 1. PMID 26598391
- [Result] Cagnazzo F, Mantilla D, Rouchaud A, Brinjikji W, Lefevre PH, Dargazanli C, Gascou G, Riquelme C, Perrini P, di Carlo D, Bonafe A, Costalat V. Endovascular Treatment of Very Large and Giant Intracranial Aneurysms: Comparison between Reconstructive and Deconstructive Techniques-A Meta-Analysis. AJNR Am J Neuroradiol. 2018 May;39(5):852-858. doi: 10.3174/ajnr.A5591. Epub 2018 Mar 15. PMID 29545248